CLINICAL TRIAL: NCT02818777
Title: A Randomized, Double Blind, Placebo-controlled Crossover Study of Tolerability and Efficacy of Cannabidiol (CBD) on Tremor in Parkinson's Disease
Brief Title: A Study of Tolerability and Efficacy of Cannabidiol on Tremor in Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Colorado Department of Public Health and Environment (Other Government); GW Research Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-0929
Record Dates: First submitted 2016-05-06; First posted 2016-06-30 (Estimated); Results first posted 2019-02-19 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2019-01

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; Tremor; tolerability; safety; cognition; anxiety; psychosis; mood; dyskinesia; cannabidiol; cannabis; efficacy; sleep; motor symptoms; non-motor symptoms; quality of life; marijuana
MeSH Terms: conditions — Parkinson Disease; Tremor; Anxiety Disorders; Psychotic Disorders; Dyskinesias; Marijuana Abuse | interventions — Cannabidiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- cannabidiol (Experimental): GWP42003-P oral solution, is purified cannabidiol (purity of ≥98%, 100 mg/ml cannabidiol in sesame oil with anhydrous ethanol with added sweetener (sucralose) and strawberry flavoring).
  Started at 5 mg/kg/day and is increased by 2.5-5 mg/kg at 3-5 day intervals to a target dose of 20 mg/kg/day.
  Interventions: Drug: cannabidiol

INTERVENTIONS:
Drug: cannabidiol — Purified CBD, is a strawberry flavored liquid, in sesame oil, provided as 100 mg/ml, extracted from high CBD plant material.
  A component of cannabis that has evidence suggesting it is relatively safe and perhaps neuroprotective, reduces tremor, anxiety and psychosis and is well tolerated in PD. Besides limiting the psychoactive effect of THC, studies support that CBD has anti-inflammatory, anticonvulsant, anti-oxidant, anxiolytic and antipsychotic properties.
  Other Names: GWP42003-P

SUMMARY:
The major purpose of the Stage 1 is to study the safety and tolerability of the proposed dosage regimen of the study drug. The form of cannabidiol (CBD) used in this study is GWP42003, supplied by GW Pharmaceuticals. The dosage regime is based on their experience. This is an open label study in 10 subjects, during which the dose is gradually increased to the manufacturers recommended target dose, with tolerability being evaluated at each dose level. Based on the response of subjects in the Stage 1, a target dose is determined for the next stage. Standardized tools will be administered to study both tolerability and efficacy. Efficacy assessments are simply explorative, and are done to look for an effect that warrants specific or different evaluation in the next stage.

DETAILED DESCRIPTION:
Persons with Parkinson's disease (PD) have progressive disabling tremor, slowness, stiffness, balance impairment, cognitive deficits, psychiatric symptoms, autonomic dysfunction, fatigue and insomnia. Tremor may interfere with necessary daily and work functions. The disorder affects approximately seven million people globally. The total economic cost in the US is around 23 billion dollars. In addition to economic costs, PD reduces quality of life of those affected and their caregivers.

Cognitive impairment is a common feature and ranges from delayed recall in early stages to global dementia in up to 80% at end stage. PD with dementia has been associated with reduced quality of life, shortened survival, and increased caregiver distress.

Depression, anxiety and psychosis are also common and are particularly disabling in PD, even at the earliest stages. These symptoms have important consequences for quality of life and daily functioning, are associated with increased carer burden and risk for nursing home admission. Anxiety affects up to 40% of patients with PD, and may predate motor symptoms by several years. The most common anxiety disorders in PD are panic attacks (often during off-periods), generalized anxiety disorder, and simple and social phobias. Psychotic symptoms vary in frequency according to the definition used. If mild forms are included, these affect up to 50% of patients. Visual hallucinations are the most common type. However, hallucinations occur in all sensory domains and delusions of various types are also relatively common. The impact of psychosis is substantial in that it is associated with dementia, depression, earlier mortality, greater caregiver strain, and nursing home placement.

Current therapies are inadequate. Medications have improved the prognosis of PD, but also have problematic adverse effects. Since treatment of PD is often unsatisfactory and since marijuana has recently become legal and readily available in Colorado, persons with PD have been trying it. Patients have heard from the internet, support groups and other sources that marijuana is helpful. Most are doing so on their own, without the supervision or even knowledge of their neurologist. In a survey conducted in the spring of 2014 in University of Colorado Movement Disorders Center (UCMDC) clinic about 5% of 207 PD patients, average age 69, reported using marijuana. In the same clinic, about 30% of the PD patients have asked doctors during their visits over the past 6 months about marijuana. In another study Katerina Venderova and colleagues reported that 25% of PD patients had taken cannabis in the General University Hospital in Prague.

PD mostly affects the elderly, and with the cognitive, psychiatric and motor problems, subjects are prone to falls. Cannabis is well documented to cause psychosis, slowness, and incoordination. Studies have also shown that chronic users have structural and functional CNS alterations. Thus cannabis is expected to be risky in persons with PD. Further, there are many components of cannabis, and the cannabis preparations being sold in Colorado vary widely in composition. There are no definitive data regarding the benefits and risks of these various preparations in PD. Studies on safety and efficacy are greatly needed to protect this fragile Colorado population.

Cannabidiol (CBD) is a cannabinoid that is present to a lesser extent in street marijuana, and limits delta-9-tetrahydrocannabinol (THC)'s psychoactive effect. CBD acts in some experimental models as an anti-inflammatory, anticonvulsant, anti-oxidant, anti-emetic, anxiolytic and antipsychotic agent, and therefore has potential beneficial medical uses. Further, animal studies suggest that CBD is neuroprotective, perhaps due to reported anti-oxidative and anti-inflammatory actions.

Human trials report that CBD decreases anxiety and causes sedation in healthy individuals, decreases psychotic symptoms in schizophrenia and PD, and improves motor and non-motor symptoms and alleviates levodopa-induced dyskinesia in PD. The ratio of THC to CBD plays a role in the preparation's therapeutic outcome: strains of cannabis with higher concentrations of CBD did not produce short-term memory impairment vs. strains with higher concentrations of THC and lower concentrations of CBD.

Many clinicians who suspect cannabis may have a positive effective upon a particular patient group have no idea of the cannabinoid profile that is being used. Without knowing the composition, it is impossible to draw any conclusions simply because of the huge variety of strains utilised.

Given the current literature regarding CBD: possible neuroprotective effect, good tolerability, anxiolytic and antipsychotic effects and general lack of be well tolerated in PD, including its effect on tremor, the investigators hypothesize that CBD would be well tolerated and would reduce tremor, anxiety and psychosis, and would stabilize cognitive decline in PD. First the investigators will perform an open label study to determine a reasonable dose, and then a randomized, double-blind, placebo-controlled crossover study to evaluate the efficacy and tolerability of oral CBD on tremor and other important aspects of PD. A strength of the study is that it uses well defined form or CBD.

Stage 1: Open Label Dose Escalation Tolerability Study

Primary Specific Aim: To confirm that the dosage regimen of CBD, in the form of GWP42003-P recommended by the study drug manufacturer is safe and tolerated in 10 subjects with PD. GWP42003-P is started at 5 mg/kg/day and is increased by 5 mg/kg at 3 day intervals to a target dose of 25 mg/kg/day.

Secondary Specific Aim: To examine the effect of CBD on severity & duration of tremor and other conditions that are problematic in PD.

The dose escalation tolerability study will be conducted in 10 subjects (the investigators will be recruiting up to 15 subjects to end up with 10) as an open label study lasting approximately 3 weeks followed by a 2-week safety follow up. Subjects are closely monitored as the dose is titrated. Subjects will have a screening visit, a baseline visit within the next three weeks, a visit when subjects are on 20 mg/kg/day, a final assessment visit when subjects have been on the maximal tolerated or the targeted dose for 10-15 days, and a safety visit 2 weeks later. The subject is to be on the maximal tolerated or targeted dose for 10-15 days. Subjects will be called on the 3rd day of each dose. During phone calls subjects are monitored for adverse events, especially excessive daytime sleepiness, symptoms of hepatotoxicity, as well as changes in medical history and concomitant medications. Subjects are also called 3 days after stopping the study drug to check for signs of withdrawal.

ELIGIBILITY:
Stage 1:

Inclusion criteria:

* Male or female subjects between 45 and 78 years of age inclusive.
* Willing and able to give informed consent.
* Idiopathic PD, per UK Parkinson's Disease Society (UKPDS) Brain Bank Clinical Diagnostic Criteria
* Rest tremor amplitude score of ≥2 in any limb on question 3.17 of the MDS-UPDRS (ON state).
* Anti-parkinsonian medication is fixed for at least 1 month prior to study entry
* If MoCA<22 subject must have a legally authorized representative (LAR) sign the consent, and must have a designated caregiver that agrees to ensure study protocols followed. This includes accompanying patient to study visits and being available for study phone calls.
* Must have a driver to drive them to and from study visits
* Has a significant other (someone who knows the subject well) that is appropriate for doing the NPI assessment, can accompany patient to study visits, and agrees to do so
* Agrees to not take more than 1 gram per day of acetaminophen, due to a possible interaction with study drug that could increase risk of hepatotoxicity.

Exclusion criteria:

* Known or suspected allergy to cannabinoids or excipients used in the study drug formulation.
* Cannabinoids taken currently or in the previous 30 days.
* History of drug or alcohol dependence; defined by prior inpatient stay(s) for this or that patient stats s/he has a history of this.
* Use of dopamine blockers within 180 days and amphetamine, cocaine, and MAO-A inhibitors within 90 days of baseline.
* Currently taking tolcapone, valproic acid, felbamate, niacin, isoniazid and ketoconazole due to risk of liver injury and clobazam and ketoconazole because of risk of toxic interactions with the study drug. These medications need to be stopped 90 days before the baseline visit.
* Unstable medical condition.
* Any of the following laboratory test results at screening:

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maureen A Leehey, M.D., Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado School of Medicine, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cannabidiol: GWP42003-P oral solution, is purified cannabidiol (purity of ≥98%, 100 mg/ml cannabidiol in sesame oil with anhydrous ethanol with added sweetener (sucralose) and strawberry flavoring).
  Started at 5 mg/kg/day and is increased by 2.5-5 mg/kg at 3-5 day intervals to a target dose of 20 mg/kg/day.
  cannabidiol: Purified CBD, is a strawberry flavored liquid, in sesame oil, provided as 100 mg/ml, extracted from high CBD plant material.
  A component of cannabis that has evidence suggesting it is relatively safe and perhaps neuroprotective, reduces tremor, anxiety and psychosis and is well tolerated in PD. Besides limiting the psychoactive effect of THC, studies support that CBD has anti-inflammatory, anticonvulsant, anti-oxidant, anxiolytic and antipsychotic properties.
Period: Overall Study
Arm/Group | Cannabidiol
Started | 13 (The number of baseline participants was 13.)
Completed | 10
Not Completed | 3
Not completed — Adverse Event | 3

BASELINE CHARACTERISTICS:
Arm/Group | Cannabidiol
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.15 (6.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Severity of Participants Reporting Study-related Adverse Events at Each Dose Level
Description: Severity of each specific adverse event was scored as 0=no adverse event, 1=mild adverse event, 2=moderate adverse event, and 3=sever adverse event. The range of severity is 0-3. Higher scores mean a worse outcome. The severity was expressed as mean (standard deviation).
Time Frame: Every 3rd day on each dose level, assessed up to 5 weeks
Population: 13 PD patients were included in safety analysis group because they were all treated with study drug.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Cannabidiol 5 mg/kg/Day: GWP42003-P oral solution, is purified cannabidiol (purity of ≥98%, 100 mg/ml cannabidiol in sesame oil with anhydrous ethanol with added sweetener (sucralose) and strawberry flavoring).
  Dosage: 5 mg/kg/day cannabidiol: Purified CBD, is a strawberry flavored liquid, in sesame oil, provided as 100 mg/ml, extracted from high CBD plant material.
  A component of cannabis that has evidence suggesting it is relatively safe and perhaps neuroprotective, reduces tremor, anxiety and psychosis and is well tolerated in PD. Besides limiting the psychoactive effect of THC, studies support that CBD has anti-inflammatory, anticonvulsant, anti-oxidant, anxiolytic and antipsychotic properties.
- Cannabidiol 7.5 mg/kg/Day: GWP42003-P oral solution, is purified cannabidiol (purity of ≥98%, 100 mg/ml cannabidiol in sesame oil with anhydrous ethanol with added sweetener (sucralose) and strawberry flavoring).
  Dosage: 7.5 mg/kg/day cannabidiol: Purified CBD, is a strawberry flavored liquid, in sesame oil, provided as 100 mg/ml, extracted from high CBD plant material.
  A component of cannabis that has evidence suggesting it is relatively safe and perhaps neuroprotective, reduces tremor, anxiety and psychosis and is well tolerated in PD. Besides limiting the psychoactive effect of THC, studies support that CBD has anti-inflammatory, anticonvulsant, anti-oxidant, anxiolytic and antipsychotic properties.
- Cannabidiol 10 mg/kg/Day: GWP42003-P oral solution, is purified cannabidiol (purity of ≥98%, 100 mg/ml cannabidiol in sesame oil with anhydrous ethanol with added sweetener (sucralose) and strawberry flavoring).
  Dosage: 10 mg/kg/day cannabidiol: Purified CBD, is a strawberry flavored liquid, in sesame oil, provided as 100 mg/ml, extracted from high CBD plant material.
  A component of cannabis that has evidence suggesting it is relatively safe and perhaps neuroprotective, reduces tremor, anxiety and psychosis and is well tolerated in PD. Besides limiting the psychoactive effect of THC, studies support that CBD has anti-inflammatory, anticonvulsant, anti-oxidant, anxiolytic and antipsychotic properties.
- Cannabidiol 15 mg/kg/Day: GWP42003-P oral solution, is purified cannabidiol (purity of ≥98%, 100 mg/ml cannabidiol in sesame oil with anhydrous ethanol with added sweetener (sucralose) and strawberry flavoring).
  Dosage: 15 mg/kg/day cannabidiol: Purified CBD, is a strawberry flavored liquid, in sesame oil, provided as 100 mg/ml, extracted from high CBD plant material.
  A component of cannabis that has evidence suggesting it is relatively safe and perhaps neuroprotective, reduces tremor, anxiety and psychosis and is well tolerated in PD. Besides limiting the psychoactive effect of THC, studies support that CBD has anti-inflammatory, anticonvulsant, anti-oxidant, anxiolytic and antipsychotic properties.
- Cannabidiol 20 mg/kg/Day: GWP42003-P oral solution, is purified cannabidiol (purity of ≥98%, 100 mg/ml cannabidiol in sesame oil with anhydrous ethanol with added sweetener (sucralose) and strawberry flavoring).
  Dosage: 20 mg/kg/day cannabidiol: Purified CBD, is a strawberry flavored liquid, in sesame oil, provided as 100 mg/ml, extracted from high CBD plant material.
  A component of cannabis that has evidence suggesting it is relatively safe and perhaps neuroprotective, reduces tremor, anxiety and psychosis and is well tolerated in PD. Besides limiting the psychoactive effect of THC, studies support that CBD has anti-inflammatory, anticonvulsant, anti-oxidant, anxiolytic and antipsychotic properties.
- Cannabidiol 25 mg/kg/Day: GWP42003-P oral solution, is purified cannabidiol (purity of ≥98%, 100 mg/ml cannabidiol in sesame oil with anhydrous ethanol with added sweetener (sucralose) and strawberry flavoring).
  Dosage: 25 mg/kg/day cannabidiol: Purified CBD, is a strawberry flavored liquid, in sesame oil, provided as 100 mg/ml, extracted from high CBD plant material.
  A component of cannabis that has evidence suggesting it is relatively safe and perhaps neuroprotective, reduces tremor, anxiety and psychosis and is well tolerated in PD. Besides limiting the psychoactive effect of THC, studies support that CBD has anti-inflammatory, anticonvulsant, anti-oxidant, anxiolytic and antipsychotic properties.
Arm/Group | Cannabidiol 5 mg/kg/Day | Cannabidiol 7.5 mg/kg/Day | Cannabidiol 10 mg/kg/Day | Cannabidiol 15 mg/kg/Day | Cannabidiol 20 mg/kg/Day | Cannabidiol 25 mg/kg/Day
Number analyzed (Participants) | 13 | 8 | 12 | 10 | 8 | 3
units on a scale
  Somnolence | 1 (0) | 1 (0) | 1 (0) | 1.25 (0.5) | 1.143 (0.345) | 1.25 (0.5)
  Fatigue | 1 (0) | 1 (0) | 1 (0) | 1.667 (0.577) | 1.25 (0.5) | 1 (0)
  Weight gain | 1.333 (0.577) | 0 (0) | 1 (0) | 1 (0) | 1 (0) | 0 (0)
  increased appetite | 1 (0) | 0 (0) | 0 (0) | 1 (0) | 0 (0) | 0 (0)
  Diarrhea | 1 (0) | 1 (0) | 1 (0) | 1.667 (0.842) | 1 (0) | 1.4 (0.775)
  Weight loss | 0 (0) | 1 (0) | 0 (0) | 1 (0) | 0 (0) | 0 (0)
  Abdominal pain | 0 (0) | 0 (0) | 1 (0) | 1 (0) | 0 (0) | 1 (0)
  Nausea | 0 (0) | 0 (0) | 1 (0) | 2 (0) | 1 (0) | 0 (0)
  Diziness | 0 (0) | 0 (0) | 1 (0) | 1 (0) | 1 (0) | 0 (0)
  Weakness | 0 (0) | 0 (0) | 1 (0) | 2 (0) | 0 (0) | 0 (0)
  Anorexia | 0 (0) | 0 (0) | 0 (0) | 2 (0) | 0 (0) | 2 (0)
  Vomiting | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (0) | 0 (0)
  Fever | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (0)

2. Primary Outcome: Number of Participants Had Changes in Orthostatic Blood Pressure
Description: Orthostatic blood pressure will be monitored at each study visit.
Time Frame: Baseline and 5 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Cannabidiol
Number analyzed (Participants) | 13
Participants | 0

3. Primary Outcome: Number of Participants Had Changes in Physical Exam
Description: A physical exam will be performed at each study visit.
Time Frame: Baseline and 5 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Cannabidiol
Number analyzed (Participants) | 13
Participants | 0

4. Primary Outcome: Number of Participants Had Changes in EKG
Description: EKG will be performed at each study visit.
Time Frame: Baseline and 5 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Cannabidiol
Number analyzed (Participants) | 13
Participants | 0

5. Primary Outcome: Number of Participants Had Changes in Laboratory Values
Description: Laboratory tests (hematology, serum chemistry, and urinalysis) will be evaluated at each study visit.
Time Frame: Baseline and 5 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Cannabidiol
Number analyzed (Participants) | 13
Participants | 5

6. Primary Outcome: Proportion of Subjects That Drop Out of the Study Due to Study Drug Intolerance
Description: Assessing the proportion of subjects that drop out of the study due to study drug intolerance.
Time Frame: Baseline and 5 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Cannabidiol
Number analyzed (Participants) | 13
Participants | 3

7. Primary Outcome: Change in Movement Disorder Society-Unified Parkinsons Disease Rating Scale Total Score
Description: There are four parts: Part I (Non-motor experiences of daily living, scores range 0-52), Part II (motor experiences of daily living, scores range 0-52), Part III (motor examination, scores range 0-132) and Part IV (motor complications scores range 0-24). Subscales are summed to a total score, ranging 0-260. Higher scores mean a worse outcome.
Time Frame: Baseline and 5 weeks
Population: 10 Participants completed the study drug treatment and were included in the efficacy analysis group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cannabidiol
Number analyzed (Participants) | 10
score on a scale | -7.70 (9.393)

8. Primary Outcome: Change in Montreal Cognitive Assessment (MoCA)
Description: MoCA - is designed as a rapid screening instrument for mild cognitive dysfunction. It assesses different cognitive domains: attention and concentration, executive functions, memory, language, visual -constructional skills, conceptual thinking, calculation. Scores range 0-30. Higher values represent a better outcome.
Time Frame: Baseline and 5 weeks
Population: 10 Participants completed the study drug treatment and were included in efficacy analysis group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cannabidiol
Number analyzed (Participants) | 10
score on a scale | 1.0 (1.491)

9. Primary Outcome: Change in Anxiety Short Form
Description: This includes 8 items that assess severity of anxiety. Scores range 8-40. Higher values represent a worse outcome.
Time Frame: Baseline and 5 weeks
Population: 10 participants completed the study drug treatment and were included in efficacy analysis group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cannabidiol
Number analyzed (Participants) | 10
score on a scale | 0.33 (3.5668)

10. Primary Outcome: Change in Neuropsychiatric Inventory (NPI)
Description: Assessing neuropsychiatric symptoms and psychopathology of patients with Alzheimer's disease and other neurodegenerative disorders. It has proven to be sensitive to change and has been employed to capture treatment related behavioral.Total NPI scores range 0-120. Higher values represent a worse outcome.
Time Frame: Baseline and 5 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cannabidiol
Number analyzed (Participants) | 10
score on a scale | -0.125 (1.5526)

11. Primary Outcome: Change in Depression Short Form
Description: This includes 8 items that assess severity of depression. Score range 8-40. Higher values represent a worse outcome.
Time Frame: Baseline and 5 weeks
Population: 10 Participants completed the study drug treatment and were included in the efficacy analysis group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cannabidiol
Number analyzed (Participants) | 10
score on a scale | -0.85 (3.132)

12. Primary Outcome: Change in Scales for Outcomes in Parkinson's Disease (SCOPA)-Sleep-night Time Sleep
Description: A valid, reliable, short scale that is used to evaluate night time sleep problems in PD. Scores range 0-18. Higher values represent a worse outcome.
Time Frame: Baseline and 5 weeks
Population: 10 Participants completed the study drug treatment and were included in the efficacy analysis group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cannabidiol
Number analyzed (Participants) | 10
score on a scale | -2.80 (3.91)

13. Primary Outcome: Change From Baseline of REM Sleep Behavior Disorder Screening Questionnaire (RBDSQ)
Description: 10-item, patient self-rating instrument assessing the subject's sleep behavior with short questions that have to be answered by either "yes" or "no". Scores range 0-13. Higher values represent a worse outcome.
Time Frame: Baseline and 5 weeks
Population: 10 Participants completed the study drug treatment and were included in the efficacy analysis group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cannabidiol
Number analyzed (Participants) | 10
score on a scale | -0.7 (1.767)

14. Primary Outcome: Change in Emotional and Behavioral Dyscontrol Short Form
Description: 8 items that assess severity of emotional and behavioral dyscontrol. Scores range 8-40. Higher values represent a worse outcome.
Time Frame: Baseline and 5 weeks
Population: 10 Participants completed the study drug treatment and were included in the efficacy analysis group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cannabidiol
Number analyzed (Participants) | 10
score on a scale | -4.69 (6.144)

15. Primary Outcome: Change in Pain Severity Form
Description: This will assess severity of pain. Scores range 3-15. Higher scores represent a worse outcome.
Time Frame: Baseline and 5 weeks
Population: 10 Participants completed the study drug treatment and were included in the efficacy analysis group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cannabidiol
Number analyzed (Participants) | 10
score on a scale | -1.86 (4.711)

16. Primary Outcome: Change in Questionnaire for Impulsive-Compulsive Disorders in Parkinson's Disease-Rating Scale (QUIP-RS)
Description: To measure severity of symptoms and support a diagnosis of impulse control disorders and related disorders in PD. Total QUIP-RS scores were summed by 6 subscores (gambling 0-16, Sex 0-16, Buying 0-16, Eating 0-16, Hobbyism-punding 0-32, and PD Medication use 0-16), range 0-112. Higher scores represent a worse outcome.
Time Frame: Baseline and 5 weeks
Population: 10 Participants completed the study drug treatment and were included in the efficacy analysis group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cannabidiol
Number analyzed (Participants) | 10
score on a scale | 0 (0)

17. Primary Outcome: Change in Fatigue Severity Scale
Description: A self-report 9-item questionnaire with questions related to how fatigue interferes with certain activities and rates its severity. Scores range 9-63. Higher values represent a worse outcome.
Time Frame: Baseline and 5 weeks
Population: 10 Participants completed the study drug treatment and were included in the efficacy analysis group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cannabidiol
Number analyzed (Participants) | 10
score on a scale | -0.5 (11.4625)

18. Primary Outcome: Change in International Restless Legs Syndrome Study Group Rating Scale for Restless
Description: This encompasses a ten-question instrument for measuring severity of restless legs syndrome (RLS). Score range 0-40. Higher values represent a worse outcome.
Time Frame: Baseline and 5 weeks
Population: 10 Participants completed the study drug treatment and were included in the efficacy analysis group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cannabidiol
Number analyzed (Participants) | 10
score on a scale | -1.2 (4.517)

19. Primary Outcome: Change in Unified Dyskinesia Rating Scale (UDysRS)
Description: To evaluate involuntary movements often associated with treated Parkinson's disease. Total UDysRS scores is the sum of historical sub-scores (0-60) and objective sub-score (0-44). Total scores range 0-104. Higher values represent a worse outcome.
Time Frame: Baseline and 5 weeks
Population: 10 Participants completed the study drug treatment and were included in the efficacy analysis group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cannabidiol
Number analyzed (Participants) | 10
score on a scale | 1.0 (3.887)

20. Secondary Outcome: Change in MDS-UPDRS Tremor Score (Total of Items 3.17 and 3.18) in the ON State
Description: Sum of items 3.17 and 3.18 of Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) evaluates the rest tremor amplitude (3.17, score range 0-20) and constancy of rest tremor (3.18 score range 0-4). The sum scores of 3.17 and 3.18 range 0-24. Higher values represent a worse outcome.
Time Frame: Baseline and 5 weeks
Population: 10 Participants completed the study drug treatment and were included in the efficacy analysis group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cannabidiol
Number analyzed (Participants) | 10
score on a scale | -0.4 (1.2649)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Cannabidiol
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 13/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cannabidiol (N=13)
Diarrhea (Gastrointestinal disorders) | 11
Somnolence (Nervous system disorders) | 9
Fatigue (General disorders) | 8
Weight gain (Metabolism and nutrition disorders) | 4
Abdominal pain (Gastrointestinal disorders) | 3
Dizziness (Nervous system disorders) | 3
weight loss (Metabolism and nutrition disorders) | 2
nausea (Gastrointestinal disorders) | 2
anorexia (Gastrointestinal disorders) | 2
increased appetite (Gastrointestinal disorders) | 2
headache (Nervous system disorders) | 2
vomiting (Gastrointestinal disorders) | 1
flatulence (Gastrointestinal disorders) | 1
gastroesophageal reflux (Gastrointestinal disorders) | 1
allergic reaction (Skin and subcutaneous tissue disorders) | 1
spasm (Musculoskeletal and connective tissue disorders) | 1
fever (General disorders) | 1
weakness (Nervous system disorders) | 1
Elevated liver function tests (Hepatobiliary disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-12): https://cdn.clinicaltrials.gov/large-docs/77/NCT02818777/Prot_SAP_000.pdf